CLINICAL TRIAL: NCT06621654
Title: A Randomized, Partially Blinded, Positively Controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine in a Population Aged 2 Months and Older
Brief Title: Clinical Trial of Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CTP-DHMCV-003
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-08

CONDITIONS: Haemophilus Influenzae Type B Infection
Keywords: Vaccine; Safety; Immunogenicity; 2 months of age and older
MeSH Terms: conditions — Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Experimental vaccine group 1A (Experimental): Subjects aged 18-59 years
  Interventions: Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine
- Experimental vaccine group 2A (Experimental): Subjects aged 1-5 years
  Interventions: Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine
- Control vaccine group 2B (Active Comparator): Subjects aged 1-5 years
  Interventions: Biological: Haemophilus Influenzae Type b Conjugate Vaccine
- Experimental vaccine group 3A (Experimental): Subjects aged 6-11 months
  Interventions: Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine
- Control vaccine group 3B (Active Comparator): Subjects aged 6-11 months
  Interventions: Biological: Haemophilus Influenzae Type b Conjugate Vaccine
- Experimental vaccine group 4A (Experimental): Subjects aged 2 months
  Interventions: Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine
- Control vaccine group 4B (Active Comparator): Subjects aged 2 months
  Interventions: Biological: Haemophilus Influenzae Type b Conjugate Vaccine

INTERVENTIONS:
Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine — 1 dose (0.5ml) of vaccine on day 0, Intramuscular injection
  Arms: Experimental vaccine group 1A
Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine — 1 dose (0.5ml) of vaccine on day 0, Intramuscular injection
  Arms: Experimental vaccine group 2A
Biological: Haemophilus Influenzae Type b Conjugate Vaccine — 1 dose (0.5ml) of vaccine on day 0, Intramuscular injection
  Arms: Control vaccine group 2B
Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine — 3 doses (0.5ml per dose) at day 0, 1 month, and 18 months of age, Intramuscular injection
  Arms: Experimental vaccine group 3A
Biological: Haemophilus Influenzae Type b Conjugate Vaccine — 3 doses (0.5ml per dose) at day 0, 1 month, and 18 months of age, Intramuscular injection
  Arms: Control vaccine group 3B
Biological: Lyophilized Haemophilus Influenzae Type b Conjugate Vaccine — 4 doses (0.5ml per dose) at day 0, 2, 4 month, and 18 months of age, Intramuscular injection
  Arms: Experimental vaccine group 4A
Biological: Haemophilus Influenzae Type b Conjugate Vaccine — 4 doses (0.5ml per dose) at day 0, 2, 4 month, and 18 months of age. Intramuscular injection
  Arms: Control vaccine group 4B

SUMMARY:
This trial is a randomized, partially blinded, positively controlled phase I clinical study. A total of 160 persons aged 18-59 years, 1-5 years, 6-11 months and 2 months (60-89 days) will be recruited into the trial, and the enrollment will be done according to the progression of age groups, from the oldest to the youngest, and the initial safety assessment will be conducted on the 8th day after the first dose of vaccination for each age group, and the next group will be enrolled only after the safety is confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 2 months, 6-11 months, 1-5 years, and 18-59 years at the time of screening
* Informed consent is obtained from the subject and the subject and/or guardian (attorney-in-fact) is able to sign the informed consent form
* Subjects are able and willing to comply with the requirements of the clinical trial protocol and are able to complete the full study follow up

Exclusion criteria for first dose:

* 2 months old, 6 months old ~ 5 years old people have been vaccinated with Hib-containing vaccines
* 2-month-old, 6~11-month-old infants who were born prematurely (delivered before the 37th week of gestation), low birth weight (birth weight <2500g)
* 2-month-old, 6~11-month-old infants with abnormal labor and delivery, history of asphyxia rescue, history of neurological damage
* Those with history of Haemophilus influenzae type b infection
* Those with history of epilepsy, convulsions, convulsions, cerebral palsy, or history of psychiatric illness or family history or other progressive neurological diseases
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), or other autoimmune diseases
* History of allergy to vaccines or vaccine components, severe side effects to vaccines such as urticaria, dyspnea, angioneurotic edema
* Female with positive urine pregnancy test or breastfeeding subjects, subjects or their partners with pregnancy plan within 6 months (only for 18~59 years old)
* Fever with axillary temperature > 37.0°C
* Known or suspected to be suffering from acute diseases or serious chronic diseases (including: serious respiratory diseases, serious cardiovascular diseases, liver and kidney diseases, serious skin diseases, malignant tumors, tuberculosis, etc.); or in the acute exacerbation of chronic diseases
* Those who have hypertension that cannot be controlled by medication (at the time of on-site measurement: systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥100 mmHg) (only applicable to 18~59 years old)
* Any of the routine blood biochemistry indexes during the screening period judged to be clinically significant by the investigator (only applicable to 2~5, 18~59 years old)
* Have no spleen or functional absence of spleen
* Suffering from thrombocytopenia, bleeding disorders, or other coagulation disorders (which may cause contraindication to intramuscular injection)
* Immunosuppressive therapy, anti-allergy therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, surface corticosteroids for acute uncomplicated dermatitis) within the past 6 months
* Received blood products within 3 months prior to receiving the experimental drug
* Participation in other studies involving interventional studies within 1 month prior to receiving the investigational drug and/or during the study participation period
* Having received an injectable live attenuated vaccine within 14 days or another vaccine within 7 days prior to vaccination
* In the judgment of the investigator, due to a variety of medical, psychological, social or other conditions that are contrary to the trial protocol or that affect the subject's ability to sign informed consent

Exclusion criteria for subsequent doses

* A vaccine-related serious adverse event occurred after the previous dose of vaccination
* Who has experienced a Grade 3 or higher allergic reaction related to the vaccine after the previous dose of vaccination
* Any other factors that, in the judgment of the investigator, make the subject unsuitable for continued participation in the clinical trial

Ages: 2 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adverse reactions in all subjects | Within 30 days of each dose of vaccine

SECONDARY OUTCOMES:
Adverse reactions in all subjects | Within 30 minutes of each dose of vaccine
Adverse events in all subjects | Within 30 days of each dose of vaccine
Incidence of SAEs in all subjects | From the first dose to 6 months after full vaccination
Incidence of abnormal and clinically significant (CS) white blood cell counts, hemoglobin, platelet counts, Alanine aminoTransferase (ALT), Aspartate Transaminase (AST), and TBIL assays in subjects 18-59, 2-5 years of age | Day 8 post-immunization
Proportion of 2-month-old subjects with anti-Hib-PRP antibody concentrations ≥1.0 μg/ml | 30 days after basic immunization, before booster immunization, 30 days after booster immunization
Positive transfer rate of anti-Hib-PRP antibodies in 2-month-old subjects | 30 days after basic immunization, before booster immunization, 30 days after booster immunization
Positivity of anti-Hib-PRP antibodies in 2-month-old subjects | 30 days after basic immunization, before booster immunization, 30 days after booster immunization
Geometric Mean Concentration (GMC) of anti-Hib-PRP antibodies in 2-month-old subjects | 30 days after basic immunization, before booster immunization, 30 days after booster immunization
Geometric Mean Increase (GMI) of anti-Hib-PRP antibodies in 2-month-old subjects | 30 days after basic immunization, before booster immunization, 30 days after booster immunization

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Li, Principal Investigator — Chongqing Center for Disease Control and Prevention (Chongqing Academy of Preventive Medicine)
Locations (1):
- Jiulongpo District Center for Disease Control and Prevention, Chongqing, China